CLINICAL TRIAL: NCT05857267
Title: Phase IV, Multicenter, Double-blind, Randomized, Controlled, Parallel-group, Trial to Evaluate the Efficacy and Safety of Dozolamide 2%/Timolol 0,5% PF vs Dorzolamide 2%/Timolol 0,5% BAK-preserved in OAG or OH
Brief Title: Dorzolamide+Timolol Multidose Preservative-free vs Dorzolamida+Timolol BAK Preserved Efficacy and Safety
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorios Poen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANTIGLAULC01
Record Dates: First submitted 2023-03-30; First posted 2023-05-12 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — dorzolamide; dorzolamide-timolol combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dorzolamide+Timolol PF (Experimental): Glaucotensil TD LC, Laboratorios Poen
  Interventions: Drug: Dorzolamide / Timolol Ophthalmic Solution
- Dorzolamide + Timolol BAK (Experimental): Glaucotensil TD, Laboratorios Poen
  Interventions: Drug: dorzolamide/timolol

INTERVENTIONS:
Drug: Dorzolamide / Timolol Ophthalmic Solution — Dorzolamide-timolol fixed combination in a preservative-free multidose device
  Other Names: Glaucotensil TD LC
  Arms: Dorzolamide+Timolol PF
Drug: dorzolamide/timolol — Dorzolamide-timolol BAK-preserved fixed combination
  Other Names: Glaucotensil TD
  Arms: Dorzolamide + Timolol BAK

SUMMARY:
The goal of this study is to evaluate the tolerability of the new formulation of Dorzolamide+Timolol preservative free developed in OSD Aptar Pharma multidose system in comparison with Dorzolamide +Timolol BAK preserved ophthalmic formulation.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* Patients with POAG and OH
* PIO < 20 mmHg
* Under treatment with Dorzolamide + Timolol BAK preserved at least 6 month after
* OSDI > 13 & one of these ocular signs (BUT <6sec or Schirmer test < 5 mm/5min or corneal staining positive)
* Corneal thickness between 520-580 um.

Exclusion Criteria:

* Patient with severe respiratory diseases (asthma, COPD and other bronchospactic diseases).
* Patient with cardiovascular diseases (Sinus Bradycardia, AV Block, Cardiac Failure, Cardiogenic Shock).
* Severe renal impairment (CrCl <30 mL/min)
* Progressive diseases of the retina other than glaucoma
* Inflammation and/or infecctions active
* Ocular surface syndrome other than Ocular Surface disease
* Eyelid disorder
* Systemic adminsitration of Betablockers or carbonic anhydrase inhibitors
* Patient that requires another antigluacomatous eye drop other than fixed combination of Dorzolamide/Timolol
* Patients who use regularly lubricant eye drops
* Patient who use regularly contact lenses
* Patient with autoinmune diseases
* Patients who underwent kerato-refractive laser procedures, cornea or corneal surface surgery, including, but not limited to, LASIK and PRK, within 6 months prior to the baseline visit.
* Patients who have undergone a laser procedure or intraocular surgery or extraocular in either eye within 6 months prior to the baseline visit.
* Patients with severe central visual field loss in either eye based onclinical judgment of the investigator. For the Humphrey and Octopus perimeters, the severe loss The visual field is defined as a sensitivity less than or equal to 10 dB in at least two(2) of the four (4) visual field test points closest to the fixation point
* Patients with known hypersensitivity to any of the components of bothdrugs under study.
* Pregnant or lactating women.
* Women of childbearing age who are not using a contraceptive method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Symptoms | Change from baseline in OSDI score at 24 weeks
  OSDI questtionarie

SECONDARY OUTCOMES:
Intraocular preassure | Change from baseline in PIO (mmHg) at 24 weeks
  Intraocular preassure (PIO) by GAT
Break-up Time | Change from baseline BUT (seconds) at 24 weeks
  Break-up Time (BUT)
SCHIRMER-ITEST | Change from baseline Shirmer test (mm) at 24 weeks
  Schirmer test without anesthesia
Conjunctival Hyperemia | Change from baseline in porcentaje of patients with conjunctival hyperemia at 24 weeks
  Conjunctival Hyperemia
Satisfaction questionnaire | Change from baseline of patient satisfaction at 24 weeks using a 5-point likert scale
  Satisfaction questionnaire
Best corrected visual acuity | Change from baseline visual acuity at 24 weeks
  snellen scale 20/20
Treatment preference | Treatment preference with respect previous treatment at Week 24
  Treatment preference

OTHER OUTCOMES:
Superficial corneal epithelium density | Change from baseline superficial corneal epithelium density at 48 weeks
  Superficial corneal epithelium density analyzed by confocal microscopy expresed by cells /mm2
Basal corneal epithelium density | Change from baseline basal corneal epithelium density at 48 weeks
  Basal corneal epithelium density analyzed by confocal microscopy expresed by cells /mm2
Corneal Estroma reflectivity | Change from baseline in the grade of corneal estroma reflectivity at 48 weeks specify by 4 grade scale reported by Martone et al. .
  Corneal Estroma reflectivity analyzed by confocal microscopy expresed by 5-point scale of grade
Corneal nerve density | Change from baseline corneal nerve density at 48 weeks
  Corneal nerve density analyzed by confocal microscopy expresed by cells /mm2
Neuroma density | Change from baseline neuroma density at 48 weeks
  Neuroma density analyzed by confocal microscopy expresed by neuromas/mm2
Dendrite density | Change from baseline dendrite density at 48 weeks
  Dendrite density analyzed by confocal microscopy expresed by dendrites/mm2
Corneal nerve tortuosity | Change from baseline in the grade of corneal nerve tortousity at 48 weeksusing a 5 point scale reported by Oliviera-Soto et al.
  Corneal nerve tortuosity analyzed by confocal microscopy expresed by 5-point scale of grade
Endothelial cell density | Change from baseline endothelial cell count at 48 weeks
  endothelial cell density analyzed by confocal microscopy expresed by cells/mm2
Conjuctival epithelium density | Change from baseline conjuctival epithelium density at 48 weeks
  Conjuntival epithelium density analyzed by confocal microscopy expresed by cells/mm2
Goblett cell density | Change from baseline goblett cell density at 48 weeks
  Goblett cell density nalyzed by confocal microscopy expresed by cells/mm2
Inflamatory infiltrates | Change from baseline in inflamatory infiltrates at 48 weeks
  Description of presence or absence of inflamtory cells on conjuntiva

CONTACTS AND LOCATIONS:
Locations (6):
- Argentina (6):
  - Clínica de Ojos Dr. Nano, Olivos, Buenos Aires
  - Consultorio Dr. Peyret, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Gonella Oftalmólogos, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Centro Diagnóstico Dr. Gentile, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Centro oftalmológico Dr. Casiraghi & asociados, Ciudad Autónoma de Buenos Aire, Buenos Aires F.D.
  - Consultorios de Oftalmología, Buenos Aires